CLINICAL TRIAL: NCT01961778
Title: Prospective Randomized Trial Comparing Radiofrequency Ablation and Cryotherapy for the Treatment of Barrett's Esophagus With High-Grade Dysplasia and/or Early Adenocarcinoma
Brief Title: Comparison of Treatments for Barrett's Esophagus With High-Grade Dysplasia/Early Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Norman Nishioka, MD, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013P001776
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Radiofrequency Ablation; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radio-Frequency Ablation (Active Comparator): Patients in this arm will receive treatment with radio-frequency ablation.
  Interventions: Device: Radio-Frequency Ablation
- Cryothearpy (Active Comparator): Patients in this arm will receive treatment with cryotherapy.
  Interventions: Device: Cryotherapy

INTERVENTIONS:
Device: Radio-Frequency Ablation
  Other Names: Barrx
  Arms: Radio-Frequency Ablation
Device: Cryotherapy
  Other Names: Trufreeze, CSA Medical
  Arms: Cryothearpy

SUMMARY:
Prospective randomized study comparing radiofrequency ablation and cryotherapy for the endoscopic treatment of Barrett's esophagus. The study is powered to assess clinical equivalence (non-inferior) of the treatment regimens.

DETAILED DESCRIPTION:
Adult patients found to be suitable candidates for endoscopic treatment of Barrett's esophagus (BE) with high-grade dysplasia (HGD) and/or early adenocarcinoma of the esophagus will be asked to participate in this study. Patients will be randomized to receive either radiofrequency ablation or cryotherapy. All treatments will be performed using standard MGH GI Unit protocol. A total of fifty subjects will be enrolled.

Patients who have contraindications to endoscopic treatment (e.g., bleeding diathesis, pregnancy, severe medical comorbidities, advanced liver disease) or who decline participation in the study will be ineligible. Patients unable to provide their own consent will also be excluded.

This is a single-site study to be conducted at MGH.

After obtaining written informed consent, the patient will be randomized to receive either radiofrequency ablation or cryotherapy. Treatments will be carried out in accordance with standard MGH GI Unit practice. The primary endpoint of the study is the percentage of Barrett's esophagus ablated at the first follow-up visit (typically 2-3 months following therapy). At this point, the patient's role in the study will be terminated. They will continue to receive routine follow-up by their physician as needed.

ELIGIBILITY:
Inclusion Criteria:

* suitable candidates for endoscopic treatment of Barrett's esophagus (BE) with high-grade dysplasia (HGD) and/or early adenocarcinoma of the esophagus

Exclusion Criteria:

* contraindications to endoscopic treatment (e.g., bleeding diathesis, pregnancy, severe medical comorbidities, advanced liver disease)
* refusal to participate in the study

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Barrett's esophagus ablated during the initial treatment session. | 2-3 months
  The primary endpoint of this study is the percentage of Barrett's esophagus ablated during the initial treatment session.

SECONDARY OUTCOMES:
Patient discomfort | 2-3 days
  The degree of patient discomfort (pain, amount of narcotics used) will be assessed during a telephone call to the patient 24-48 hours following the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Norman S Nishioka, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States